CLINICAL TRIAL: NCT07149428
Title: Longitudinal Deep Phenotyping of Central Mechanisms in Dysosmia: A Pilot Study Using Electrobulbogram (EBG), Functional MRI (fMRI), and Diffusion-Weighted Imaging (DWI)
Status: Not yet recruiting | Type: Observational
Sponsor: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002331; 002331-DC
Record Dates: First submitted 2025-08-29; First posted 2025-09-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01-20

CONDITIONS: Respiratory Tract Infection; Smell Disorder; Influenza; Rhinosinusitis; COVID-19; Depression; Parosmia; Hyposomia; Normosomia; Anosmia
Keywords: SMELL; Chemotherapy; chemicals; Mood; Diet; Neuroimaging; electrobulbogram; fMRI; Cognition; Toxins
MeSH Terms: conditions — Respiratory Tract Infections; Olfaction Disorders; Influenza, Human; Rhinosinusitis; COVID-19; Depression; Anosmia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Anosmia: participants with complete loss of smell
- Hyposmia: participants with reduced smell sensitivity
- Normosmia (Healthy control cohort): participants with normal smell function
- Parosmia: participants with a distorted smell perception

SUMMARY:
Background:

Loss of the sense of smell can seriously affect a person's quality of life. The ability to smell can be damaged by many factors, including illnesses, injuries, and exposure to toxic chemicals. The effects can vary, including complete loss of smell, partial loss, and parosomia, which is when things smell differently than they should.

Objective:

To study how brain function changes in people with different types of smell disorders. Also, to look at how smell loss affects quality of life over time.

Eligibility:

People aged 18 years or older with a disorder that affects their sense of smell. Healthy volunteers are also needed.

Design:

Participants will have 5 study visits over 1 year. They will have various tests and procedures:

Smell tests. They will have several tests that involve smelling different items and answering questions.

Questionnaires. They will answer questions about their health, mood, sense of smell, and daily habits.

Magnetic resonance imaging (MRI) scans. They will lie on a bed that slides into a tube. Padding will hold their head still. They will smell different odors while in the scanner.

Electrobulbogram (EBG). They will wear a soft cap with sensors that measure brain activity. They will smell different odors while wearing the cap.

Nasal endoscopy. A flexible tube will be inserted into a nostril to view the inside of the nose.

Biopsy. A numbing substance will be sprayed into the nose. Then a scissor-like tool will be used to collect a sample of tissue from one or both nasal passages.

Samples of blood, urine, and nasal fluid will be taken.

DETAILED DESCRIPTION:
Study Description:

This pilot study investigates the mechanisms of parosmia, a qualitative olfactory dysfunction increasingly seen after COVID-19, by examining functional and structural brain changes and peripheral inflammation. Using neuroimaging and biochemical analysis, it aims to distinguish parosmia from other olfactory disorders and provide a foundation for future diagnostic and therapeutic approaches.

Objectives:

Primary objective:

* Evaluate the feasibility, validity, and methodological framework for deep phenotyping of acquired chemosensory disorders.
* Examine task-based functional connectivity patterns from the olfactory bulb to higher-order central processing regions across groups with varying olfactory symptoms.
* Associate central findings with peripheral inflammatory patterns at the olfactory mucosa.

Secondary Objective:

-Investigate the differences and longitudinal changes in white matter microstructural integrity associated with the progression and recovery of olfactory dysfunctions across the recruited patient population.

Tertiary objective:

-Investigate the psychophysiological impacts of altered smell perception, with an emphasis on its negative effects on dietary habits, oral health, and cognitive functions.

Endpoints:

Co-Primary Endpoints:

To identify functional connectivity differences across subgroups, with focus on parosmia. The study hypothesizes that parosmia patients exhibit neuroinflammation at the olfactory bulb or in the amygdala and hippocampus, leading to distorted valence perception. Altered connectivity between primary and secondary olfactory cortices is expected, differing significantly from hyposmia and, to a lesser extent, anosmia. These connectivity changes are expected to correlate with variations in smell function to uncover disrupted neural pathways underlying parosmia.

To identify local inflammatory signatures at the olfactory mucosa that are associated with chemosensory dysfunction and altered functional connectivity.

Secondary Endpoints:

To evaluate whether changes in functional connectivity are associated with structural alterations, specifically reduced axonal myelination between primary and secondary olfactory cortices (amygdala and hippocampus), in parosmia patients (along with their symptoms graph) compared to healthy controls and, to a lesser extent, anosmia patients. Longitudinal analysis will determine if these structural changes lead to higher-order neural degeneration or other significant brain alterations.

Tertiary endpoints:

To investigate whether regions with structural and functional differences correlate with the duration and severity of smell loss, and to assess the impact of prolonged smell dysfunction on psychological health, eating behaviors, oral health, and quality of life.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet all the following criteria:

1. Adult subjects, any sex, aged 18 or older.
2. Ability to understand and willingness to sign a written informed consent document.
3. Willingness and ability to comply with and participate in all study procedures and availability for the duration of the study.
4. Due to the extensive questionnaires (administered in English language only) that participants must complete independently, fluency in the English language is needed. Hence, participants must be able to read and understand English.

   * To maintain consistency in the study, we will prioritize enrolling individuals who have experienced olfactory loss for no more than one year. However, the duration of olfactory dysfunction can vary significantly, often due to delayed awareness or recognition of the condition. For instance, anosmia and hyposmia are frequently reported as long-term consequences of infections, meaning some participants may have experienced prolonged dysfunction. Given this variability, we will treat the duration of olfactory loss as a potential confounding factor in our data analysis, ensuring that its influence is appropriately accounted for when interpreting the results. Other than healthy controls, participants reporting smell loss must also meet one or more of the following criteria to be eligible for the study:

<!-- -->

1. General Smell Loss:

   Individuals who have experienced any degree of smell loss or olfactory dysfunction, regardless of the cause. This includes both partial, complete to distorted loss of the sense of smell (hyposmia, anosmia or parosmia).
2. Post-COVID-19 or Virus-Related Smell Loss:

   Individuals experiencing olfactory dysfunction due to COVID-19, influenza or other respiratory viruses, leading to both acute and long-term (chronic) smell loss
3. Sinonasal Smell Loss:

   Participants diagnosed with smell loss related to sinonasal conditions, such as:
   * Chronic Rhinosinusitis: Long-term inflammation of the sinuses that impairs olfactory function.
   * Nasal Polyps: Growths in the nasal passage that obstruct airflow and affect the sense of smell.
4. Exposure to Toxic Chemicals:

Patients who have encountered olfactory dysfunction due to exposure to harmful chemicals or environmental toxins that can impair the olfactory receptors or neural pathways responsible for the sense of smell.

5. Chemotherapy-Induced Smell Loss:

Individuals who have experienced smell loss as a side effect of undergoing chemotherapy. This includes patients who are in active treatment as well as those who have completed chemotherapy but continue to suffer from olfactory impairment.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Compromised cognitive ability: Including dementia, intellectual disability, or severe learning disorders, traumatic brain injury,
2. Major psychotic and neurological condition: Examples include schizophrenia, bipolar disorder, Parkinson's disease, and multiple sclerosis, epilepsy.
3. Normosmia (healthy) controls must not have:

   -Any history of smell or taste loss.

   -Prior nasal surgery.
   * Acute or chronic olfactory disorders.
4. Diagnosis of depression or anxiety.
5. None of the participants should be current smokers or consume drugs such as cocaine, heroin, opioids, or marijuana.
6. Pregnancy

   * Participants who report moderate depressive symptoms (BDI >= 20) but do not have a formal diagnosis of depression will not be automatically excluded from the study. Instead, their responses will be flagged for clinical review and referral. If, upon follow-up, a clinical diagnosis of depression is confirmed, they may be excluded in accordance with the study's exclusion criteria. Participants who indicate any level of suicidality on question 9 will be evaluated on a case-by-case basis. If there is any indication of risk, they will be referred for immediate clinical evaluation. Depending on the outcome and the risk level determined, a decision will be made regarding their continued participation, with participant safety as the highest priority.

fMRI-Specific Exclusion Criteria

-Metallic implants, such as pacemakers, cochlear implants, or orthopedic devices, can pose safety risks during an MRI scan due to the strong magnetic fields used in the procedure. These implants can also cause artifacts in the MRI images, distorting the data and making it difficult to obtain accurate results.

* Non-removable piercings can also cause safety risks and image artifacts during MRI scans. These piercings may heat up or move in response to the magnetic fields, potentially causing injury or discomfort to the participant.
* Permanent makeup and tattoos, particularly those containing metallic pigments, can pose risks during MRI due to the potential for heating or movement of the pigments. These effects can cause discomfort or burns and will also create artifacts in the MRI images.
* Pregnancy is an exclusion criterion for MRI studies due to the potential risks to the fetus from the strong magnetic fields and radiofrequency energy used in the procedure. Additionally, pregnant participants will find it uncomfortable to lie still in the MRI machine for extended periods, which could affect the quality of the images.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will enroll adults aged 18 and older who are fluent in English and able to provide informed consent and comply with study procedures. Participants will include both healthy volunteers with normal smell and individuals with olfactory dysfunction of varying causes, such as post viral (including COVID-19), sinonasal disease, chemical exposure, or chemotherapy-related smell loss. To maintain consistency, preference will be given to participants who have experienced smell loss within the past year, through those with longer durations of dysfunction may be included.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-10-14 (Estimated)

PRIMARY OUTCOMES:
Functional Connectivity Differences in Olfactory Dysfunction | baseline, 3, 6, 9 and 12 months
  differences in functional brain connectivity between parosmia, anosmia and hyposmia groups, assessed longitudinally.

SECONDARY OUTCOMES:
Structural Brain Changes in Olfactory Dysfunction | baseline, 3, 6, 9 and 12 months
  Structural brain architecture differences in olfactory-related regions, measured with neuroimaging.
Cognitive, Mood and Dietary Impact of Olfactory Dysfunction | baseline, 3, 6, 9 and 12 months
  Associations between olfactory function and changes in cognition, depressive symptoms and dietary habits, evaluated through surveys and behavioral measures.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Levy, M.D., Principal Investigator — National Institute on Deafness and Other Communication Disorders (NIDCD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_002331-DC.html